CLINICAL TRIAL: NCT02134678
Title: Assessing Change in Short Term Therapy for Depression Using ESM
Brief Title: Assessing Change in Short Term Therapy for Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Greensboro (Other)
Responsible Party: Principal Investigator, Kari M Eddington, Assistant Professor, University of North Carolina, Greensboro
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1R21MH090414-01A1 (NIH)
Record Dates: First submitted 2014-05-05; First posted 2014-05-09 (Estimated); Last update posted 2015-05-01 (Estimated); Status verified 2015-04

CONDITIONS: Depression
Keywords: self-system therapy; cognitive therapy; depression; psychotherapy; mechanisms of action
MeSH Terms: conditions — Depression | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- self-system therapy (Experimental): self-system therapy for depression
  Interventions: Behavioral: self-system therapy
- cognitive therapy (Active Comparator): cognitive therapy for depression
  Interventions: Behavioral: cognitive therapy

INTERVENTIONS:
Behavioral: self-system therapy
  Arms: self-system therapy
Behavioral: cognitive therapy
  Arms: cognitive therapy

SUMMARY:
This study will compare mechanisms of action in two forms of brief psychotherapy for major depressive disorder in adults. A treatment that targets deficits in motivation in depression is expected to show greater improvements in motivation and pursuit of personal goals compared to a second treatment that targets irrational thoughts that are typical in depression.

DETAILED DESCRIPTION:
Outcome studies have shown that several forms of psychotherapy are effective for depression, but questions about how, why, and when these treatments work remain. The proposed study answers the call for innovative research designs that allow for more intensive, individualized data collection that can address complex questions about the dynamic nature of treatment-related change. In this R21 application, we propose a proof-of-concept study using an innovative application of experience sampling methodology (ESM) that combines the idiographic advantages of single-subject research with the statistical advantages associated with larger samples and multilevel analyses. ESM involves sampling aspects of behavior occurring in the participant's everyday environment, thereby enhancing ecological validity and reducing retrospective bias. Thirtyfour adults with primary major depressive disorder will be randomly assigned to 16 weeks of either selfsystem therapy (SST), a new short-term, empirically-supported psychotherapy for depression that targets deficits in incentive motivation and goal pursuit, or treatment-as-usual (TAU). Participants will complete a battery of individual difference and diagnostic measures at pretreatment. One week of intensive ESM will be collected at both pre- and post-treatment, during which participants will be signaled at random times during each day to answer questions about current functioning in several domains (e.g., affect, cognition, and goal pursuit) delivered via a phone-based interactive voice response (IVR) system. Throughout the 16 weeks of treatment, participants will complete similar IVR assessments on two randomly-selected days per week. The proposed study will test three main hypotheses. (1) Patients in SST will show greater increases in engagement with promotion goals and activities as well as greater increases in goal-related daily experiences of positive affect over the course of treatment compared to patients in TAU. (2) Patients in SST will show greater decreases in engagement with prevention goals and activities as well as greater decreases in goal- related daily experiences of negative affect over the course of treatment compared to patients in TAU. (3) Within the SST condition, a history of failure to pursue or achieve promotion goals and individual differences in chronic regulatory orientation (i.e., strength of orientation toward promotion and prevention goals) will moderate the effects of SST on changes in depressive symptoms and on daily experiences of promotion goal engagement. The proposed research will have a significant impact on an important public health problem and will expand our knowledge of how psychotherapy for depression works. The data to be obtained from this study will provide a sound empirical and theoretical framework for largerscale programmatic research on the nature of treatment-induced change processes in patients with depression.

ELIGIBILITY:
Inclusion Criteria:

* primary diagnoses of major depressive disorder or dysthymia
* age 18-60

Exclusion Criteria:

* bipolar
* substance abuse
* acute suicidality
* antisocial or borderline personality disorder
* cognitive impairment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2011-05; Primary Completion 2014-05 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Change in Depressive symptoms - Beck Depression Inventory-II | post-treatment and 6 month follow up

SECONDARY OUTCOMES:
Change in Anxiety - Beck Anxiety Inventory | post-treatment and 6 month follow up

CONTACTS AND LOCATIONS:
Locations (1):
- UNC Greensboro, Greensboro, North Carolina, United States

REFERENCES:
- [Derived] Eddington KM, Silvia PJ, Foxworth TE, Hoet A, Kwapil TR. Motivational deficits differentially predict improvement in a randomized trial of self-system therapy for depression. J Consult Clin Psychol. 2015 Jun;83(3):602-616. doi: 10.1037/a0039058. Epub 2015 Apr 13. PMID 25867448